CLINICAL TRIAL: NCT00867555
Title: Effects of the Green Tea Extract TEAVIGO High in EGCG, on Postprandial Fat Oxidation in Overweight Volunteers
Brief Title: Green Tea, High in Epigallocatechin Gallate (EGCG) and Postprandial Fat Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Ellen E Blaak, Prof, Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: MEC 08-3-052
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGCG (Experimental): Double blind randomized, placebo-controlled cross-over design with two arms:
  * the green tea extract TEAVIGO, high in EGCG and
  * placebo
  Interventions: Dietary Supplement: Effect of the green tea extract TEAVIGO, high in EGCG, on postprandial fat oxidation
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Effect of the green tea extract TEAVIGO, high in EGCG, on postprandial fat oxidation

INTERVENTIONS:
Dietary Supplement: Effect of the green tea extract TEAVIGO, high in EGCG, on postprandial fat oxidation — green tea extract TEAVIGO, high in EGCG

SUMMARY:
The body of evidence regarding the health benefits of green tea has grown considerably during the last decade and includes antioxidant properties, anti- cancer, anti-obesity and anti-diabetes effects. There has been evidence that green tea extract favorably affect body weight and body fat and has positive effects on blood glucose control

Aim of this study is to investigate the short term effect (3-day)of TEAVIGO (high in the catechin EGCG) on postprandial fat oxidation during different phases of the postprandial period in overweight subjects. Secondly, in a subset of volunteers changes in lipolysis and glucose metabolism will be studied in skeletal muscle and adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 50 y
* BMI 25.0-29.9 kg/m2
* Normal fasting glucose <6.1 mmol/L
* Blood pressure (systolic blood pressure 100-150 mmHg, diastolic blood pressure 60-90 mmHg)
* Weight stable in last 3 months (±2 kg)

Exclusion Criteria:

* pregnant, lactating or (post)menopausal women
* regular smokers
* people with intensive fitness training eg athletes
* habitual consumption of green or black tea (more than 1 or 2 cups a day, respectively)
* not more than 300 mg/day caffeine consumption

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
postprandial fat oxidation | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, PhD, Prof, Principal Investigator — Maastricht University
Locations (1):
- Dept Human Biology, Maastricht University, Maastricht, Netherlands